CLINICAL TRIAL: NCT07159256
Title: The Effect of Information Processing Speed on Motor Function, Balance, Gait, and Quality of Life in Patients With Ischemic Stroke
Brief Title: Impact of Processing Speed on Motor, Balance, Gait, and Quality of Life in Stroke"
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Dudu Kübra AKYOL, Principal Investigator, Istanbul Aydın University
Other Study IDs: IstanbulIAU
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Ischaemic Stroke
Keywords: Information Processing Speed; Motor Function; Balance; Gait; Quality of Life; ischaemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: All participants will be patients diagnosed with first-ever ischemic stroke, aged 40 years or older, hemodynamically stable, literate, and without pre-stroke psychiatric, neurological, visual, auditory, or orthopedic conditions that could affect mobilization. Participants will undergo a series of standardized assessments including information processing speed (Symbol Digit Modalities Test), motor function (Fugl-Meyer Assessment), balance (Berg Balance Scale and Sense4Motion Euleria Health device), gait (Timed Up and Go Test), and quality of life (Stroke-Specific Quality of Life Scale). The aim is to evaluate the relationship between processing speed and functional outcomes in ischemic stroke rehabilitation.

SUMMARY:
Stroke rehabilitation programs are traditionally designed based on the evaluation of motor and sensory impairments starting from the acute phase. Although studies in diseases such as multiple sclerosis and Parkinson's disease have shown that information processing speed may affect motor function and balance, no such study has been conducted in stroke patients.

This study aims to investigate the effect of information processing speed on motor function, balance, gait, and quality of life in patients with ischemic stroke.

DETAILED DESCRIPTION:
A review of the literature reveals that in stroke patients, motor and sensory impairments are evaluated beginning in the acute phase, and rehabilitation programs are structured accordingly. While research has demonstrated that information processing speed can influence motor function and balance in other neurological conditions such as multiple sclerosis and Parkinson's disease, no similar studies exist for stroke populations.

The investigators hypothesize that early evaluation of motor, sensory, and cognitive deficits in patients with ischemic stroke, and incorporating these findings into rehabilitation programs, may positively impact prognosis.

This study will recruit patients admitted for treatment at the Physical Medicine and Rehabilitation Unit of Istanbul Aydın University VM Medical Park Florya Hospital. Inclusion criteria are: age ≥ 40 years, first-ever ischemic stroke, hemodynamic stability, literacy, and absence of pre-stroke psychiatric, neurological, visual, auditory, or orthopedic conditions that may affect mobilization. Additionally, patients must score full points in the vision and speech domains of the NIHSS after stroke.

Eligible participants' demographic and clinical data will be recorded. Information processing speed will be assessed using the Symbol Digit Modalities Test (SDMT). Motor function will be evaluated with the Fugl-Meyer Assessment (FMA), balance with the Berg Balance Scale (BBS) and the Sense4Motion Euleria Health device, gait with the Timed Up and Go Test (TUG), and quality of life with the Stroke-Specific Quality of Life Scale (SS-QOL).

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* First-ever ischemic stroke
* Hemodynamically stable
* Able to read and write (literate)
* No history of psychiatric, neurological, visual, auditory, or orthopedic conditions prior to stroke that could affect mobilization
* After stroke, full scores in the vision and speech domains according to the NIH Stroke Scale (NIHSS)

Exclusion Criteria:

* Recurrent stroke
* Post-stroke visual or hearing impairment
* Neglect
* Aphasia
* Conditions causing impaired consciousness such as dementia, confusion, or delirium
* Presence of cardiovascular or orthopedic conditions after stroke that prevent mobilization
* Age 75 years or older

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 40-74 years who experienced a first-ever ischemic stroke and are hemodynamically stable. Eligible participants will be literate, without prior psychiatric, neurological, visual, auditory, or orthopedic conditions affecting mobilization. Patients must have full scores in the vision and speech domains of the NIH Stroke Scale (NIHSS) after stroke. Individuals with recurrent stroke, severe cognitive or language impairments, post-stroke visual or auditory deficits, neglect, cardiovascular or orthopedic conditions preventing mobilization, or those aged 75 years and older will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-10-07 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) Score | At baseline (single assessment)
  The Symbol Digit Modalities Test (SDMT) will be used to assess information processing speed. The test requires participants to match symbols with corresponding numbers according to a reference key within 90 seconds. The total number of correct responses will be recorded, with higher scores indicating better processing speed.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) Score | At baseline (single assessment)
  The Berg Balance Scale (BBS) will be used to evaluate functional balance. The test consists of 14 tasks, including sitting, standing, reaching, and turning activities, each scored on a 5-point scale from 0 (unable to perform) to 4 (independent performance). The total score ranges from 0 to 56, with higher scores indicating better balance.
Fugl-Meyer Assessment (FMA) Score | At baseline (single assessment)
  The Fugl-Meyer Assessment (FMA) will be used to evaluate motor function in stroke patients. The scale assesses movement, coordination, and reflexes of the upper and lower extremities. Scores range from 0 to 100, with higher scores indicating better motor function and recovery.
Stroke-Specific Quality of Life Scale (SS-QOL) Score | At baseline (single assessment)
  The Stroke-Specific Quality of Life Scale (SS-QOL) will be used to assess health-related quality of life. It consists of 49 items across 12 domains (e.g., mobility, mood, energy, self-care, social roles). Each item is scored on a 5-point Likert scale, with higher scores indicating better quality of life.
Balance Assessment with Sense4Motion Euleria Health / Euleria Lab Device | At baseline (single assessment)
  The Sense4Motion Euleria Health (Euleria Lab) device will be used for objective balance assessment. This wearable inertial sensor system measures postural stability and body sway during standardized balance tasks. Quantitative parameters such as sway velocity, sway area, and stability index will be recorded. Lower sway values and higher stability indices indicate better balance performance.
Timed Up and Go Test (TUG) with Euleria Health / Euleria Lab | At baseline (single assessment)
  The gait module of Euleria Health (Euleria Lab) device will be used to perform the Timed Up and Go (TUG) test. Participants will be asked to rise from a chair, walk three meters, turn, return, and sit down. The device's inertial sensors will record spatiotemporal gait parameters such as duration (seconds), number of steps, gait speed, and turning characteristics. Lower times and more stable gait parameters indicate better functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan ÖZKOÇAK, MD, Study Chair — Istanbul Aydın University; Özden Erkan Oğul, Asst. Prof, Study Chair — Medipol University; İbrahim H Ural, MD, Study Chair — Beykent University; Arzu DİNÇ YAVAŞ, MD, Study Chair — Istanbul Aydın University; Dudu K AKYOL, PT, Principal Investigator — Istanbul Aydın University
Locations (1):
- Istanbul Aydın University, Istanbul, Küçükçekmece, Turkey (Türkiye)